CLINICAL TRIAL: NCT02740400
Title: Endobronchial Ultrasonography With a Guide Sheath Versus Computed Tomography-guided Transthoracic Needle Biopsy in the Diagnosis of Peripheral Pulmonary Lesions
Brief Title: A Comparison Between EBUS-GS and CT-guided Lung Biopsy in Diagnosis of Peripheral Pulmonary Lesions.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Jun Wang, Chief director of Department of Thoracic Surgery, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CDI2014-2-4084
Record Dates: First submitted 2016-04-05; First posted 2016-04-15 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Lung Neoplasms
Keywords: Endobronchial ultrasonography; guided sheath; diagnosis; accuracy; complication
MeSH Terms: conditions — Lung Neoplasms; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CT-TTNB (Experimental): patients receive CT-TTNB to diagnose PPLs.
  Interventions: Procedure: CT-TTNB
- EBUS-GS (Experimental): patients receive EBUS-GS to diagnose PPLs.
  Interventions: Procedure: EBUS-GS

INTERVENTIONS:
Procedure: EBUS-GS — The equipment for EBUS-GS includes super-thin bronchoscope BF-P260F, endobronchial ultrasonic system EU-M30S, ultrasonic probe UM-S20-17S, and guided sheath kit K201. All facilities are provided by Olympus Co. The EBUS-GS procedure was performed by thoracic surgeons. The patient was in supine position, under general anesthesia, and provided ventilatation through laryngeal mask. First, the operator placed super-thin bronchoscope into the bronchus of interest, inserted the probe covered with GS through a work channel. Later, adjusted the bronchoscope and probe to obtain classical ultrasonic graphs. The assistant fixed the bronchoscope, pulled the probe out, and placed the brush and biopsy forceps, respectively, through the GS. This process was assisted using x-ray fluoroscope or not.
  Arms: EBUS-GS
Procedure: CT-TTNB — The devices for CT-TTNB includes Lightspeed VCT spiral CT(GE co.) and Quickcore(COOK Co.) biopsy kit. The kit includes a sheath(5cm in length and 16G in outer diameter) and a automatic biopsy needle(15cm in length and 18G in outer diameter). The patient stays in supine, prone or lateral position according to the lesion's location. The first chest CT scan is performed to confirm the location of the lesion and make an optimal entry point. Then, after sterilization and 2% lidocaine local anesthesia, the sheath is stabbed into chest wall through the entry point. The second CT scan is performed to make sure that the sheath stays in proper angle and depth. The operator places the needle through the sheath and enter the lesion. Then fire the biopsy needle and repeat the procedure twice or third time. The last CT scan is conducted to determine whether pneumothorax or hemorrhage occurred.
  Arms: CT-TTNB

SUMMARY:
This is a randomized controlled trail aiming at comparing the diagnostic value and safety of endobronchial ultrasonography with a guide sheath(EBUS-GS) and computed tomography-guided transthoracic needle biopsy(CT-TTNB) for peripheral pulmonary lesions (PPLs). Patients eligible for the inclusion criteria are diagnosed using either EBUS-GS or CT-TTNB randomly. The diagnostic indicators such as sensitivity, specificity, and accuracy are compared between the two groups. Post-procedure complications are recorded.

DETAILED DESCRIPTION:
CT-TTNB is widely used in the diagnosis of PPLs and its sensitivity for lung cancer remains as high as 90%. However, the relatively high rate of complications such as pneumothorax, hemoptysis, pulmonary hemorrhage, severe chest pain, and bad tolerance in patients limits its application.

EBUS-GS is an emerging technology, Kurimoto in 2004 performed transbronchial lung biopsy(TBLB) assisted by EBUS-GS, and the sensitivity of diagnosing lung cancer was 81%, and it was proved to be a safe procedure with very small amount of pneumothorax and hemoptysis.

Till now there is only one randomized controlled study comparing the diagnostic value of CT-TTNB and EBUS-GS; however, it did not complete the enrollment of patients on schedule. In addition, all the other studies were retrospective. Hence this prospective study was performed to determine the diagnostic value and safety of EBUS-GS and CT-TTNB for PPLs.

ELIGIBILITY:
Inclusion Criteria:

* Lesions presented as nodule or mass in CT imaging and located at the distal end of the segmental bronchus; invisible under normal bronchoscope; no pathological results were obtained before biopsy procedure; patients can tolerate video assisted thoracic surgery(VATS) lobectomy or wedge resection; all patients provided written informed consent.

Exclusion Criteria:

* Presence of central pulmonary lesion and visible under the bronchoscope; lesions presented as exudative or consolidation in CT imaging; the location was unsuitable for CT-guided biopsy; presence of pneumothorax or pleural effusion patients have contraindication for EBUS-GS or CT-TTNB,such as cardiopulmonary dysfunction, cachexia, thrombocytopenia or coagulopathy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-06 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Safety. It is measured by the incidence rate of all adverse events during or after EBUS-GS or CT-TTNB. | 30 days
  Adverse events include: 1)pneumothorax or pulmonary hemorrhage which are observed in CT scan after CT-TTNB; 2)patient's complaint of chest pain or dyspnea after returning the ward, and bedside X-ray shows pneumothorax or decreased respiratory auscultation，and drainage should be performed; 3)postoperative hemoptysis and usage of hemostatic agents;4)severe chest pain, but no pneumothorax in chest film, no T wave or ST segment changes in ECG,and analgesics should be used;5)new tumor or subcutaneous nodules are found in the needle channel during the follow-up;6)other adverse events: such as pleural reaction; arrhythmia, continuous hypoxemia or persistent hypotension during anesthesia process; hoarseness after EBUS-GS,and cricoarytenoid joint dislocation is found by laryngoscope.

SECONDARY OUTCOMES:
Diagnostic value. It is measured by the diagnostic accurate rate between the two groups. | 6 months
  If the pathological results from EBUS-GS or CT-TTNB show lung cancer, metastatic carcinoma or other malignant tumors, they are recorded as accurate.
  If the patient undergoes the following surgical treatment, the histological results from the resected tissues are "golden standard".
  If the pathological diagnosis is non-neoplastic and the patient does not receive surgery, the follow-up radiographic findings will decide. If there is no change or reduction in size, it is considered as accurate, otherwise false negative.
  If the biopsy diagnosis are mucosa, cartilage, coagulation, necrosis or other description that can not make a predisposed diagnosis. They are also recorded as negative results.

CONTACTS AND LOCATIONS:
Overall Officials: Guanchao Jiang, M.D., Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People'S Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kurimoto N, Miyazawa T, Okimasa S, Maeda A, Oiwa H, Miyazu Y, Murayama M. Endobronchial ultrasonography using a guide sheath increases the ability to diagnose peripheral pulmonary lesions endoscopically. Chest. 2004 Sep;126(3):959-65. doi: 10.1378/chest.126.3.959. PMID 15364779
- [Result] Hiraki T, Mimura H, Gobara H, Iguchi T, Fujiwara H, Sakurai J, Matsui Y, Inoue D, Toyooka S, Sano Y, Kanazawa S. CT fluoroscopy-guided biopsy of 1,000 pulmonary lesions performed with 20-gauge coaxial cutting needles: diagnostic yield and risk factors for diagnostic failure. Chest. 2009 Dec;136(6):1612-1617. doi: 10.1378/chest.09-0370. Epub 2009 May 8. PMID 19429718
- [Result] Fielding DI, Chia C, Nguyen P, Bashirzadeh F, Hundloe J, Brown IG, Steinke K. Prospective randomised trial of endobronchial ultrasound-guide sheath versus computed tomography-guided percutaneous core biopsies for peripheral lung lesions. Intern Med J. 2012 Aug;42(8):894-900. doi: 10.1111/j.1445-5994.2011.02707.x. PMID 22212110
- [Result] Wang Memoli JS, Nietert PJ, Silvestri GA. Meta-analysis of guided bronchoscopy for the evaluation of the pulmonary nodule. Chest. 2012 Aug;142(2):385-393. doi: 10.1378/chest.11-1764. PMID 21980059
- [Result] Hayama M, Izumo T, Matsumoto Y, Chavez C, Tsuchida T, Sasada S. Complications with Endobronchial Ultrasound with a Guide Sheath for the Diagnosis of Peripheral Pulmonary Lesions. Respiration. 2015;90(2):129-35. doi: 10.1159/000431383. Epub 2015 Jun 19. PMID 26112297